CLINICAL TRIAL: NCT04991324
Title: Cholecalciferol Comedication in Patients With Chronic Inflammatory Bowel Diseases (Crohn's Disease or Ulcerative Colitis) - the 5C-study
Brief Title: Cholecalciferol Comedication in IBD - the 5C-study
Acronym: 5C
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University Hospital, Basel, Switzerland (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2022-00899; NCT05624801 (obsolete NCT alias)
Record Dates: First submitted 2021-07-27; First posted 2021-08-05 (Actual); Last update posted 2024-12-24 (Actual); Status verified 2024-12

CONDITIONS: Inflammatory Bowel Diseases
MeSH Terms: conditions — Inflammatory Bowel Diseases | interventions — Cholecalciferol

STUDY DESIGN:
Intervention Model Description: Parallel Assignment Patient will be recruited by their regularly visit. Patients will be randomly assigned to be supplemented with monthly capsules (monthly group), weekly capsules (weekly group) or no supplementation (control group).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- weekly supplementation (Experimental): Weekly administration of a capsule containing 24'000 IU vitamin D, corresponding to a dose of approximately 3500 IU per day, as comedication to the usual treatment during 6 months.
  Interventions: Drug: Vitamin D3
- monthly supplementation (Active Comparator): Monthly administration of a capsule containing 24'000 IU vitamin D, corresponding to a dose of approximately 800 IU per day, as comedication to the usual treatment during 6 months.
  Interventions: Drug: Vitamin D3
- control group (No Intervention): Usual treatment without vitamin D supplementation.

INTERVENTIONS:
Drug: Vitamin D3 — 24,000 IU cholecalciferol
  Other Names: D3 VitaCaps
  Arms: monthly supplementation; weekly supplementation

SUMMARY:
Vitamin D deficiency (defined as 25(OH)-vitamin D serum level <50 nmol/ l) is associated with irritable bowel disease (IBD). National guidelines recommend the administration of 800 -4000 IU cholecalciferol daily for an effective treatment, especially during the winter (poor sun exposition). Cumulative intermittent administration monthly or weekly is possible. The study aims to compare inflammation activity (primary outcome) after monthly or weekly treatment with soft capsules containing 24'000 IU cholecalciferol compared to no vitamin D supplementation. Quantification of 25(OH)-vitamin D serum values is a secondary outcome. The investigators will use newly developed soft capsules.

DETAILED DESCRIPTION:
Monthly supplementation: Monthly administration of a capsule containing 24'000 IU vitamin D, corresponding to a dose of approximately 800 IU per day, as comedication to the usual treatment during 6 months.

Weekly supplementation: Weekly administration of a capsule containing 24'000 IU vitamin D, corresponding a dose of approximately 3500 IU per day, as comedication to the usual treatment during 6 months.

Control: Usual treatment without vitamin D supplementation. All 3 groups: In a follow-up phase of 6 months, all participants can choose whether they want a monthly vitamin D supplementation or not.

ELIGIBILITY:
Inclusion Criteria:

* diagnosis of Crohn disease or ulcerative colitis

Exclusion Criteria:

* hypercalcaemia

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Actual)
Dates: Start 2022-09-21 (Actual); Primary Completion 2024-09-15 (Actual); Study Completion 2024-09-15 (Actual)

PRIMARY OUTCOMES:
fecal calprotectin | every 2 months during 6 months
  laboratory disease activity

SECONDARY OUTCOMES:
(OH)-vitamin D serum value | every 2 months during 6 months
  serum value cholecalciferol

OTHER OUTCOMES:
disease activity score | every 2 months during 6 months
  clinical disease activity
medication adherence | every 2 months during 6 months
  adherence to vitamin D supplementation

CONTACTS AND LOCATIONS:
Overall Officials: Samuel Allemann, Prof., Study Chair — Pharmaceutical Care Research Group; Petr Hrúz, Prof., Principal Investigator — Clarunis
Locations (1):
- Clarunis, Basel, Switzerland

IPD SHARING:
Plan to Share IPD: No